CLINICAL TRIAL: NCT05889195
Title: Validation of Cxbladder Triage-Plus for the Detection of Urothelial Carcinoma in Subjects With Microscopic Hematuria (microDRIVE)
Brief Title: Detection and Risk Stratification in Veterans Presenting With Microscopic Hematuria
Acronym: microDRIVE
Status: Recruiting | Type: Observational
Sponsor: Pacific Edge Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CXB/2023/microDRIVE
Record Dates: First submitted 2023-05-22; First posted 2023-06-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-05

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial Carcinoma; microscopic hematuria; Cxbladder; Urine test; genomic test
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Cxbladder urine test — Cxbladder tests uses mRNA and DNA biomarkers in the urine to direct the management of UC from diagnosis to surveillance for disease recurrence.

SUMMARY:
It is currently debated whether the use of invasive standard of care procedures, such as cystoscopy, a procedure which involves inserting a thin camera, called a cystoscope, into the bladder to look for signs of disease, is appropriate for patients with microscopic hematuria (blood in the urine that cannot be seen with the naked eye). This is because the risk of disease (bladder cancer - urothelial carcinoma) is relatively low in this population group, approximately 3%. Invasive procedures such as cystoscopy can cause anxiety and pain, in addition to other potential side effects. This has resulted in low admittance for cystoscopy among patients with hematuria (blood in urine) in urology clinics. Therefore, there is a need for a simpler, non-invasive test that can accurately detect the presence or absence of disease (urothelial carcinoma) in patients with microscopic hematuria. Cxbladder, a non-invasive, urine-based test, has the potential to fill this role.

DETAILED DESCRIPTION:
This is a multicenter, observational study prospectively enrolling up to 1000 subjects with microscopic hematuria (three or more red blood cells per high powered field in one urinalysis; no visible blood in the urine) and gross hematuria (visible blood in urine) from US sites. This study will be conducted with subjects with a previous history of microscopic or gross hematuria referred to urology and scheduled for cystoscopy for the investigation of urothelial carcinoma. The study will aim to recruit an equal number of microscopic and gross hematuria patients, controlling the proportion of gross hematuria subjects recruited by targeting an approximate 1:1 ratio of microscopic to gross hematuria patients.

Consented, eligible subjects will undergo all standard of care tests as clinically indicated. In addition, one additional urine sample, using remote (at-home) or at-clinic sampling, will be collected to validate the performance characteristics for the Cxbladder Triage-Plus test. The urine sample collected from each subject will be a voided urine sample within 90 days prior to the scheduled cystoscopy or within 10 weeks post-cystoscopy.

The primary aim of this study is to validate the use of Cxbladder Triage-Plus as an effective diagnostic tool to:

1. Enable patients with microscopic hematuria who have a low probability of having disease (urothelial carcinoma) to be ruled out from further investigation. This could avoid expensive, invasive work-up, without compromising detection of disease.
2. Allow physicians to identify subjects at higher risk of disease (urothelial carcinoma)
3. Replace less sensitive urine-based tests (such as urine cytology or other urine genomic tests currently available)

Cxbladder results will not be reported to the subjects or the physicians. Each subject will be required to fill in the date of sample collection in the test-request form and Cxbladder tubes. The site will fill in case-report forms in a professional manner in accordance with good clinical practice (GCP).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are referred to urology and are either scheduled for a cystoscopy or have had a cystoscopic investigation within the last two months for the evaluation of hematuria meeting ONE of the following criteria:

   EITHER: (a) Microscopic hematuria, confirmed by urine microscopy of three or more RBC/HPF (or equivalent). OR: (b) Gross hematuria.
2. Physically able to provide a voided urine sample from a bladder that has not been surgically altered.
3. Able to give informed, written consent.
4. Able and willing to comply with study requirements (complete at-home urine sampling, fill in test request forms (TRFs) / tube labels and ship urine back to the central laboratory using a prepaid courier service).
5. Aged 18 years or older.

Footnotes:

1. For the microscopic hematuria patients, the recruitment priority at each respective site will be: i) Patients who have undergone initial diagnostic cystoscopy and have been scheduled for a later TURBT for suspicious lesion in the bladder. ii) Patients who are considered high risk by the AUA 2020 guidelines.
2. For gross hematuria patients, the recruitment priority at each respective site will be: i) Patients who have undergone initial diagnostic cystoscopy and have been scheduled for a later TURBT for suspicious lesion in the bladder

Exclusion Criteria:

1. Prior history of bladder malignancy.
2. Reported Cxbladder results within the last six months.
3. Prior history of upper tract urothelial carcinoma (UC) or prostatic urethral UC.
4. Reconstructed or diverted bladder (e.g., bladder augmentation, ileal conduit, Indiana pouch).
5. Subjects aged 89 years of age or older.
6. Subjects with a history of pelvic radiation.
7. Subjects currently receiving systemic chemotherapy or has had systemic chemotherapy within the last six weeks.
8. Subjects with renal failure on dialysis.
9. History of schistosomiasis.
10. Subjects who have had intervention (TURBT, diathermia, etc.,) following a previous cystoscopy.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multicenter, observational study prospectively enrolling up to 1000 subjects with microscopic hematuria (three or more red blood cells per high powered field in one urinalysis; no visible blood in the urine) and gross hematuria (visible blood in the urine) from US sites. This study will be conducted on subjects with microscopic or gross hematuria referred to urology and scheduled for cystoscopy for the investigation of urothelial carcinoma.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To validate the performance characteristics of Cxbladder Triage Plus in a US cohort which will consist of subjects with a recent history of hematuria and are referred to urology and scheduled for cystoscopy for the evaluation of hematuria. | Baseline, pre-intervention / procedure (cystoscopy): Each subject is scheduled for cystoscopy and provides one urine sample for the Cxbladder test pre-procedure
  Cxbladder Triage-Plus performance will be measured using performance characteristics such as sensitivity, specificity, negative predictive value and positive predictive value.

SECONDARY OUTCOMES:
To validate the performance characteristics and Test Negative Rate of Cxbladder Triage Plus through sub-group analysis (gross hematuria, microscopic hematuria, inflammation) for patients with a recent history of hematuria who are undergoing cystoscopy | Baseline, pre-intervention / procedure (cystoscopy): Each subject is scheduled for cystoscopy and provides one urine sample for the Cxbladder test pre-procedure
  Cxbladder Triage test performance will be measured using performance characteristics such as sensitivity, specificity, negative predictive value and positive predictive value.
To evaluate the performance characteristics of both Cxbladder Triage Plus and Cxbladder Triage in a pooled analysis with combined results generated at other clinical sites, and to the results of other published clinical studies. | Baseline, pre-intervention / procedure (cystoscopy): Each subject is scheduled for cystoscopy and provides one urine sample for the Cxbladder test pre-procedure
  Cxbladder Triage test performance will be measured using performance characteristics such as sensitivity, specificity, negative predictive value and positive predictive value.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Lough, PhD, Study Chair — Pacific Edge (Australia) Pty Ltd
Locations (4):
- United States (4):
  - Tri Valley Urology Medical Group, Murrieta, California
  - AccuMed Research Associates, Garden City, New York
  - Durham VA Health Care System, Durham, North Carolina
  - The Urology Place, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Data will be published in an anonymized report once the study is completed.